CLINICAL TRIAL: NCT06167668
Title: The Influence of Internet + Combined Family Empowerment Management Mode on Treatment Compliance of PATIENTS With CKD and the Relationship Between Psychological Status and Disease Progression
Brief Title: The Influence of Internet + Combined Family Empowerment Management Mode on Treatment Compliance of PATIENTS With CKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Jie, Associate professor, Shanxi Medical University
Other Study IDs: 2021SLL138
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Internet; Chronic Kidney Disease
Keywords: Compliance; Self-efficacy; Family empowerment management; Mental state
MeSH Terms: conditions — Renal Insufficiency, Chronic; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- combined group
  Interventions: Other: the family-centered family enabling health management mode
- traditional group
  Interventions: Other: the routine chronic disease management mode

INTERVENTIONS:
Other: the routine chronic disease management mode — indoor temperature and humidity adjustment, regular ventilation and hygiene of ward and clinic environment, promotion of patients' health awareness by distributing disease brochures, regular inspection of wards, and home nursing and health guidance based on disease knowledge when discharged
  Groups: traditional group
Other: the family-centered family enabling health management mode — The specific measures were as follows :(1) intervention group construction. (2) Online knowledge promotion. (3) Disease assessment.(4) Medication guidance reminder.(5) Enabling psychological counseling.
  Groups: combined group

SUMMARY:
To explore the effect of Internet + combined family empowerment management mode on treatment compliance of patients with chronic kidney disease (CKD) and the correlation between psychological status and disease progression.

DETAILED DESCRIPTION:
To explore the effect of Internet + combined family empowerment management mode on treatment compliance of patients with chronic kidney disease (CKD) and the correlation between psychological status and disease progression. A total of 100 patients with CKD treated in our hospital from October 2020 to October 2021 were screened and analyzed, and randomly divided into combined group and traditional group according to the number table method, with 50 patients in each group. The traditional group was implemented with the conventional chronic disease management mode, and the combined group was implemented with the Internet + combined family empowerment management mode. The differences in compliance, self-efficacy, psychological status and renal function indexes of each group were compared. Mmas-8 compliance score and GSES score showed an increasing trend. Compared with the traditional group, T2-T4MMAS-8 score and GSES score in the combined group were significantly increased with statistical differences (P < 0.05). The levels of BUN, Scr, SAS and SDS showed a decreasing trend. Compared with the traditional group, the levels of four indexes T2-T4 in the combined group were significantly decreased with statistical differences (P < 0.05). BUN, Scr were positively correlated with SAS and SDS (P< 0.05). Internet + combined family empowerment management model can effectively improve renal function, negative psychological clarity, self-efficacy and medication compliance of CKD patients, which is worthy of clinical promotion.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled subjects meet the diagnostic criteria for CKD and are confirmed to be CKD based on laboratory findings.
* After assessment, it was determined that the subject's communication was barrier-free
* No abnormal feedback was found after evaluation.
* The patient received dialysis treatment for more than 3 months, and the clinical data were complete. This is the first time they've been to the hospital.

Exclusion criteria:

* The female patient is pregnant and lactating.
* Kidney transplant patient.
* People with language communication disorders or mental diseases.
* Participants received other psychological guidance and health education interventions during the study period.

Ages: 40 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Combined with laboratory results, CKD was confirmed
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-07-24 (Estimated); Study Completion 2024-11-24 (Estimated)

PRIMARY OUTCOMES:
blood urea nitrogen | 70/5000 The four observation time points in this study were 1 day before treatment, 1 month, 3 months, and 6 months after treatment, labeled T1 to T4, respectively. T1 ~ T4 when fasting in the morning.
  5ml of fasting elbow vein was collected from patients in the morning at four study observation time points from T1 to T4, and Z206A table top medical centrifuge produced by HERMLE, Germany, was centrifuged at a speed of 1500 r/min for 0.5h to extract upper serum, which was placed in a refrigerator at -70℃ for detection.
serum creatinine | 70/5000 The four observation time points in this study were 1 day before treatment, 1 month, 3 months, and 6 months after treatment, labeled T1 to T4, respectively. T1 ~ T4 when fasting in the morning.
  5ml of fasting elbow vein was collected from patients in the morning at four study observation time points from T1 to T4, and Z206A table top medical centrifuge produced by HERMLE, Germany, was centrifuged at a speed of 1500 r/min for 0.5h to extract upper serum, which was placed in a refrigerator at -70℃ for detection.

SECONDARY OUTCOMES:
Morisky Medication Adherence Scale | Six months Max
General Self-Efficacy Scale | Six months Max
Self-Rating Anxiety Scale | Six months Max

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China